CLINICAL TRIAL: NCT02769260
Title: Comparison of Biofilm Characteristics Between an in Situ Biofilm Model of Supragingival Plaque and Natural Teeth
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Inmaculada Tomas, Senior Lecture, University of Santiago de Compostela
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pyro-Biofilm
Record Dates: First submitted 2016-04-20; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Biofilm; Dental Plaque
Keywords: pyrosequencing; 16S DNA gene; Confocal Laser Scanning Microscope; bacterial viability; bacterial diversity
MeSH Terms: conditions — Dental Plaque | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No toothbrushing during experiment and Pyrosequencing (No Intervention): Volunteers will not brush their teeth during 48 hours. Dental plaque samples will be analyse by CLSM (confocal Laser scanning microscope) and 16S DNA pyrosequencing.
- No toothbrushing during experiment (No Intervention): Volunteers will not brush their teeth during 48 hours. Dental plaque samples will be analyse by CLSM (confocal Laser scanning microscope).
- Toothbrushing during experiment (Active Comparator): 48hours-Dental plaque samples will be analyse by CLSM (confocal Laser scanning microscope).
  Interventions: Other: Toothbrushing

INTERVENTIONS:
Other: Toothbrushing — Normal toothbrushing without toothpaste or antiseptic mouthwash.
  Arms: Toothbrushing during experiment

SUMMARY:
The purpose of this study is to determine in situ the bacterial viability, thickness and bacterial diversity of a biofilm formed on different substrates in comparison to a naturally tooth-formed oral biofilm. In addition, it will be evaluated whether the restraint of oral hygiene measures may influence the development of the PL-Biofilm.

DETAILED DESCRIPTION:
* To calculate an a priori sample size, the following statistical criteria were established: an effect size of 0.35, an alpha error of 0.05 and a statistical power of 87%. Assuming these criteria and using the repeated measures ANOVA test, a sample size of 15 subjects was required.
* Bacterial viability and thickness will be analyse by Confocal Laser Scanning Microscope and Live/Dead BackLight staining solution.
* Bacterial diversity will be analyse by Pyrosequencing the 16S DNAr gene.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* good oral health status

Exclusion Criteria:

* smoker or former smoker,
* presence of dental prostheses or orthodontic devices,
* antibiotic treatment or routine use of oral antiseptics in the previous 3 months,
* presence of any systemic disease that could alter the production or composition of saliva

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Bacterial viability | Bacterial viability measured in proportion of viable/no viable bacteria after 48 hours of exposition to oral cavity
  It will be measured by analysis of images taken by Confocal laser Scanning Microscope
Bacterial diversity | Bacterial diversity measured by microbial estimators of abundance and richness after 48 hours of exposition to oral cavity
  It will be measured by 16S rDNA gene pyrosequencing and posterior bioinformatic analysis.

SECONDARY OUTCOMES:
Biofilm thickness | Oral biofilm thickness measured by analysis of sectional images after 48 hours of exposition to oral cavity
  It will be measured by analysing sectional images taken by Confocal Laser Scanning Microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Tomás Carmona, S Lecturer, Principal Investigator — Univeristy of Santiago de Compostela
Locations (1):
- Univeristy of Santiago de Compostela, Faculty of Dentistry, Santiago de Compostela, Galicia/ A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will shared in a supplementary file in the published paper